CLINICAL TRIAL: NCT04846543
Title: PMCF Study - Verification of Activa IM-Nail™ Safety and Clinical Performance
Brief Title: Bioresorbable Intramedullary Nailing of Forearm Fractures
Acronym: BRINFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Klestil (Other)
Collaborators: Bioretec Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Thomas Klestil, Univ.-Prof. DDr. Thomas Klestil, Danube University Krems
Organization: Danube University Krems (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DanubeUK3031
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Forearm Fracture
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan 1st and 2nd year (Other): Additionally to routinely follow up, there will be an MRI scan of enrolled patients after one and two years in some of the study sites
  Interventions: Other: MRI Scan

INTERVENTIONS:
Other: MRI Scan — MRI scan

SUMMARY:
The Activa IM-Nail™ is used in the fixation of forearm fractures with cast to achieve a level of reduction and stabilisation that is appropriate to the age of the child. The post-market clinical follow-up study will be performed to identify the residual risk related to re-fracture and to determine its impact to the risk/benefit ratio of Activa IM-Nail™.

DETAILED DESCRIPTION:
Residual risk related to re-fracture rate will be addressed by this PMCF study. The research question is, if the re-fracture risk with Activa IM-nail is in line with the other treatment methods, namely ESIN.

Primary objective: will be to assess clinical outcome by determining re-fracture rate of all treated patients, difference of re-fracture rate depending on the fracture type determined by X-ray (e.g. greenstick vs. non-greenstick fracture), subject's age, BMI, surgical technique, immobilization time and bony union formation.

ELIGIBILITY:
Inclusion Criteria:

* Diaphyseal forearm fractures (radius or ulna or both)
* Patients from 3 years to under 13 years, but the age limits depend on the biological development of the child and in addition

Exclusion Criteria:

* multifragmentary fractures, metaphyseal and epiphyseal fractures
* Situations where internal fixation is otherwise contraindicated, e.g., active or potential infection, or where a patient's cooperation cannot be guaranteed.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Refracture rate | First year after operation
  Assessment of refracture rate

SECONDARY OUTCOMES:
Absorption of implant | One and two years after operation
  MRI scans are performed to evaluate soft tissue reaction and biodegradability
Bony union | One year after operation
  Bony union depending on fracture type and immobilization time, return to sport
Monteggia lesion and equivalent | 2 years after operation
  Safety and performance of operative technique in Monteggia´s lesion
Cost effectiveness | 1 year after operation
  HTA assessment for different health care systems in Europe

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Roeder, MD, Principal Investigator — Landesklinikum Baden/Moedling
Locations (9):
- Landesklinikum Moedling, Mödling, Lower Austria, Austria
- Denmark (2):
  - Herlev and Gentofte University Hospital Department of Orthopedic Surgery, Herlev
  - Hvidovre Hospital, Hvidovre
- Lille University Center, Jeanne de Flandre Hospital, Lille, France
- University Medical Center Schleswig-Holstein, Campus Lübeck Department of Pediatric Surgery, Lübeck, Schleswig-Holstein, Germany
- Hungary (2):
  - Péterfy Hospital, National Trauma Center, Department of Pediatric Trauma Surgery, Budapest
  - Pécs University Hospital, Department of Pediatrics, Pécs
- Hospital Pediátrico - CHUC, EPE, Coimbra, Portugal
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korhonen L, Perhomaa M, Kyro A, Pokka T, Serlo W, Merikanto J, Sinikumpu JJ. Intramedullary nailing of forearm shaft fractures by biodegradable compared with titanium nails: Results of a prospective randomized trial in children with at least two years of follow-up. Biomaterials. 2018 Dec;185:383-392. doi: 10.1016/j.biomaterials.2018.09.011. Epub 2018 Sep 11. PMID 30292588